CLINICAL TRIAL: NCT01575756
Title: A Prospective, Controlled, Randomised, Crossover Study Investigating the Pharmacokinetic Properties, Surrogate Efficacy and Safety of Octafibrin Compared to Haemocomplettan® P/RiaSTAPTM in Patients With Congenital Fibrinogen Deficiency
Brief Title: Pharmacokinetic, Efficacy, and Safety Study of Octafibrin Compared to Haemocomplettan/Riastap
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FORMA-01
Record Dates: First submitted 2012-04-09; First posted 2012-04-11 (Estimated); Results first posted 2016-11-30 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Congenital Fibrinogen Deficiency; Afibrinogenemia
MeSH Terms: conditions — Afibrinogenemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Octafibrin followed by Haemocomplettan® P or RiaSTAPTM (Experimental): Participants received Octafibrin 70 mg/kg intravenously once followed by Haemocomplettan® P or RiaSTAPTM 70 mg/kg intravenously once 45 days later.
  Interventions: Biological: Octafibrin; Biological: Haemocomplettan® P or RiaSTAPTM
- Haemocomplettan® P or RiaSTAPTM followed by Octafibrin (Experimental): Participants received Haemocomplettan® P or RiaSTAPTM 70 mg/kg intravenously once followed by Octafibrin 70 mg/kg intravenously once 45 days later.
  Interventions: Biological: Octafibrin; Biological: Haemocomplettan® P or RiaSTAPTM

INTERVENTIONS:
Biological: Octafibrin — Octafibrin was supplied as a powder for reconstitution with water for injection.
  Other Names: Plasma derived fibrinogen concentrate
Biological: Haemocomplettan® P or RiaSTAPTM — Commercially available Haemocomplettan® P or RiaSTAPTM (same product with different names in different markets) were supplied as powders for reconstitution with water for injection.
  Other Names: Plasma derived fibrinogen concentrate

SUMMARY:
The purpose of this study is to investigate pharmacokinetic properties, surrogate efficacy and safety of Octafibrin compared to Haemocomplettan® P/RiaSTAPTM in patients with congenital fibrinogen deficiency

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years.
* Documented congenital fibrinogen deficiency (afibrinogenemia).

Exclusion Criteria:

* Life expectancy > 6 month.
* Bleeding disorder other than congenital fibrinogen deficiency.
* Presence or history of hypersensitivity to study medication.
* Presence or history of deep vein thrombosis or pulmonary embolism within 1 year prior to enrollment.
* Presence or history of arterial thrombosis with 1 year prior to enrollment.
* Hypersensitivity to human plasma products.
* Acute bleeding.
* Pregnant or currently breast-feeding women.
* Suspicion of an anti-fibrinogen inhibitor as indicated by previous in vivo recovery (if available).
* Blood or plasma donation in the 3 months prior to enrollment.
* Human immunodeficiency virus (HIV) positive with a viral load > 200 particles/µl or > 400000 copies/mL.
* End-stage liver disease.
* History of oesophageal varicose bleeding.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sigurd Knaub, PhD, Study Director — Octapharma
Locations (10):
- United States (2):
  - University of Colorado Hemophilia & Thrombosis Center, Aurora, Colorado
  - Cohen Children's Medical Center of New York, New Hyde Park, New York
- Specialized Hospital for Active Treatment "Joan Pavel", Sofia, Bulgaria
- India (3):
  - Department of Hematology St. John's Medical College Hospital, Bangalore
  - Sahyadri Speciality Hospital, Prune
  - Department of Hematology Christian Medical College, Vellore
- Iran (2):
  - Nemazee Hospital Shiraz University of Medical Sciences, Shiraz
  - Tehran University of Medical Sciences, Tehran
- Department of Hematology University Hospital, Zurich, Switzerland
- The Centre for Haemostatis and Thrombosis, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Octafibrin/FIBRYGA® Followed by Haemocomplettan® P/RiaSTAP(TM): Participants received Octafibrin/FIBRYGA® 70 mg/kg body weight (BW) intravenously once followed by Haemocomplettan® P/RiaSTAP(TM) 70 mg/kg BW intravenously once 45 days later.
- Haemocomplettan® P/RiaSTAP(TM) Followed by Octafibrin/FIBRYGA®: Participants received Haemocomplettan® P/RiaSTAP(TM) 70 mg/kg BW intravenously once followed by Octafibrin/FIBRYGA® 70 mg/kg BW intravenously once 45 days later.
Period: Treatment Period 1
Arm/Group | Octafibrin/FIBRYGA® Followed by Haemocomplettan® P/RiaSTAP(TM) | Haemocomplettan® P/RiaSTAP(TM) Followed by Octafibrin/FIBRYGA®
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | Octafibrin/FIBRYGA® Followed by Haemocomplettan® P/RiaSTAP(TM) | Haemocomplettan® P/RiaSTAP(TM) Followed by Octafibrin/FIBRYGA®
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set: All randomised participants who received at least 1 infusion of study medication (Octafibrin/FIBRYGA® and/or any part of an infusion of Haemocomplettan® P/RiaSTAP(TM)) and for whom any post-treatment data were available.
Groups:
- Full Analysis Set: All randomised participants who received at least 1 infusion of study medication (Octafibrin/FIBRYGA® and/or any part of an infusion of Haemocomplettan® P/RiaSTAP(TM)) and for whom any post-treatment data were available.
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.0 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Octafibrin/FIBRYGA® to Haemocomplettan® P/RiaSTAP(TM) for Fibrinogen Activity Normalized Area Under the Curve Unstandardized
Description: Fibrinogen activity was determined via a validated Clauss assay (fibrinogen activity) and fibrinogen-specific enzyme-linked immunosorbent assay (ie, fibrinogen antigen) using paired antibodies for fibrinogen antigen. All determinations were performed on frozen plasma samples in a central laboratory. The Clauss assay was modified and validated to achieve a limit of quantification of 0.2 g/L. The pharmacokinetic analysis was assessed individually using a non-compartmental model. Plasma levels were measured at Baseline, and at 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216, and 312 hours post-treatment. The mean ratio of normalized area under the curve was calculated as Octafibrin/FIBRYGA® over Haemocomplettan® P/RiaSTAP(TM)
Time Frame: Baseline to 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216, and 312 hours post-treatment
Population: Pharmacokinetic (PK)-per protocol dataset: All randomised participants who received ≥ 90% of the treatment (T) doses, had any post-T data, did not receive any fibrinogen (F) containing blood products between T and 14 days post-T in both study periods; had sufficient PK data for analysis; had a ≥ 50 mg/dL increase in plasma F within 4 hours post-T.
Measure: Mean (90% Confidence Interval); unit: ratio
Groups:
- Pharmacokinetic (PK)-Per Protocol Dataset: Ratio comparison of participants who received Octafibrin/FIBRYGA® 70 mg/kg body weight (BW) intravenously once, and participants who received Haemocomplettan® P/RiaSTAP(TM) 70 mg/kg BW intravenously once
Arm/Group | Pharmacokinetic (PK)-Per Protocol Dataset
Number analyzed (Participants) | 21
ratio | 1.196 [1.117 to 1.281]

2. Primary Outcome: Comparison of Maximum Clot Firmness Between Octafibrin/FIBRYGA® and Haemocomplettan® P/RiaSTAP(TM) at 1 hr Post Infusion
Description: Thromboelastometry (ROTEM®) was used to measure maximum clot firmness. Thromboelastometry is a method for the continuous measurement of clot formation. Maximum clot firmness is a functional parameter that depends on the activation of coagulation, the platelet and fibrinogen content of the blood sample, and the polymerisation and cross-linking of the fibrin network. In order to obtain comparable results from all study centres, maximum clot firmness data were assessed from frozen citrated plasma samples in a central laboratory. As these samples did not contain platelets that would be found in the whole blood assay, the fibrinogen content primarily defined the maximum clot firmness.
Time Frame: 1 hour post-treatment
Population: Full analysis set: All randomised participants who received at least 1 infusion of study medication (Octafibrin/FIBRYGA®) and/or any part of an infusion of Haemocomplettan® P/RiaSTAP(TM)) and for whom any post-treatment data were available.
Measure: Mean (95% Confidence Interval); unit: mm
Groups:
- Octafibrin/FIBRYGA®: Participants received Octafibrin/FIBRYGA® 70 mg/kg body weight (BW) intravenously once.
- Haemocomplettan® P/RiaSTAP(TM): Participants received Haemocomplettan® P/RiaSTAP(TM) 70 mg/kg BW intravenously once.
Arm/Group | Octafibrin/FIBRYGA® | Haemocomplettan® P/RiaSTAP(TM)
Number analyzed (Participants) | 22 | 22
mm | 9.68 [8.37 to 10.99] | 10.00 [8.07 to 11.93]

3. Secondary Outcome: Fibrinogen Activity Normalized Area Under the Curve Unstandardized
Description: Fibrinogen activity was determined via a validated Clauss assay (fibrinogen activity) and fibrinogen-specific enzyme-linked immunosorbent assay (ie, fibrinogen antigen) using paired antibodies for fibrinogen antigen. All determinations were performed on frozen plasma samples in a central laboratory. The Clauss assay was modified and validated to achieve a limit of quantification of 0.2 g/L. The pharmacokinetic analysis was assessed individually using a non-compartmental model. Plasma levels were measured at Baseline, and at 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216, and 312 hours post-treatment.
Time Frame: Baseline to 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216, and 312 hours post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h•kg•g/L/mg
Arm/Group | Octafibrin/FIBRYGA® | Haemocomplettan® P/RiaSTAP(TM)
Number analyzed (Participants) | 21 | 21
h•kg•g/L/mg | 1.62 (0.45) | 1.38 (0.47)

4. Secondary Outcome: Fibrinogen Activity Normalized Area Under the Curve Standardized
Description: Fibrinogen activity was determined via a validated Clauss assay (fibrinogen activity) and fibrinogen-specific enzyme-linked immunosorbent assay (ie, fibrinogen antigen) using paired antibodies for fibrinogen antigen. All determinations were performed on frozen plasma samples in a central laboratory. The Clauss assay was modified and validated to achieve a limit of quantification of 0.2 g/L. The pharmacokinetic analysis was assessed individually using a non-compartmental model. Plasma levels were measured at Baseline, and at 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216, and 312 hours post-treatment. The normalized area under the curve was standardized to a dose of 70 mg/kg.
Time Frame: Baseline to 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216, and 312 hours post-treatment
Population: Pharmacokinetic (PK)-per protocol dataset: All randomised participants who received ≥ 90% of the treatment (T) doses; had any post-T data; did not receive any fibrinogen (F) containing blood products between T and 14 days post-T in both study periods; had sufficient PK data for analysis; had a ≥ 50 mg/dL increase in plasma F within 4 hours post-T.
Measure: Mean (Standard Deviation); unit: g•h/L
Arm/Group | Octafibrin/FIBRYGA® | Haemocomplettan® P/RiaSTAP(TM)
Number analyzed (Participants) | 21 | 21
g•h/L | 113.70 (31.54) | 96.39 (32.89)

5. Secondary Outcome: Maximum Plasma Concentration Normalized (Cmaxnorm)
Description: as for outcome 3
Time Frame: Baseline to 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216, and 312 hours post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg•g/L/mg
Arm/Group | Octafibrin/FIBRYGA® | Haemocomplettan® P/RiaSTAP(TM)
Number analyzed (Participants) | 21 | 21
kg•g/L/mg | 0.018 (0.005) | 0.018 (0.005)

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) Unstandardized
Description: as for outcome 3
Time Frame: Baseline to 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216, and 312 hours post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Octafibrin/FIBRYGA® | Haemocomplettan® P/RiaSTAP(TM)
Number analyzed (Participants) | 21 | 21
g/L | 1.390 (0.369) | 1.265 (0.309)

7. Secondary Outcome: Maximum Plasma Concentration (Cmax) Standardized
Description: Fibrinogen activity was determined via a validated Clauss assay (fibrinogen activity) and fibrinogen-specific enzyme-linked immunosorbent assay (ie, fibrinogen antigen) using paired antibodies for fibrinogen antigen. All determinations were performed on frozen plasma samples in a central laboratory. The Clauss assay was modified and validated to achieve a limit of quantification of 0.2 g/L. The pharmacokinetic analysis was assessed individually using a non-compartmental model. Plasma levels were measured at Baseline, and at 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216, and 312 hours post-treatment. The maximum plasma concentration was standardized to a dose of 70 mg/kg.
Time Frame: Baseline to 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216, and 312 hours post-treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: g•h/L
Arm/Group | Octafibrin/FIBRYGA® | Haemocomplettan® P/RiaSTAP(TM)
Number analyzed (Participants) | 21 | 21
g•h/L | 1.266 (0.338) | 1.271 (0.312)

8. Secondary Outcome: Incremental in Vivo Recovery
Description: Incremental in vivo recovery was calculated as the maximum increase in plasma fibrinogen (fibrinogen activity assay data) within 4 hours post-treatment as compared with pre-treatment (expressed as an absolute mg/dL concentration in plasma), divided by the exact dose of Octafibrin/FIBRYGA® or Haemocomplettan® P/RiaSTAP(TM) (expressed as mg/kg dosed).
Time Frame: Baseline to 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216, and 312 hours post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL/(mg/kg)
Arm/Group | Octafibrin/FIBRYGA® | Haemocomplettan® P/RiaSTAP(TM)
Number analyzed (Participants) | 21 | 21
mg/dL/(mg/kg) | 1.787 (0.458) | 1.770 (0.442)

9. Secondary Outcome: Classical in Vivo Recovery
Description: Classical in vivo recovery was calculated as: 100 x the maximum increase in plasma fibrinogen (fibrinogen activity assay data) within 4 hours post-treatment as compared with pre-treatment (expressed as an absolute mg/dL concentration in plasma) x the plasma volume (mL), divided by the exact dose of Octafibrin/FIBRYGA® or Haemocomplettan® P/RiaSTAP(TM) (expressed as mg).
Time Frame: Baseline to 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216, and 312 hours post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Octafibrin/FIBRYGA® | Haemocomplettan® P/RiaSTAP(TM)
Number analyzed (Participants) | 21 | 21
percentage | 64.397 (11.519) | 66.046 (11.635)

10. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Description: as for outcome 3
Time Frame: Baseline to 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216, and 312 hours post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Octafibrin/FIBRYGA® | Haemocomplettan® P/RiaSTAP(TM)
Number analyzed (Participants) | 21 | 21
h | 2.148 (1.475) | 1.417 (2.054)

11. Secondary Outcome: Terminal Half-life (t½)
Description: as for outcome 3
Time Frame: Baseline to 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216, and 312 hours post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Octafibrin/FIBRYGA® | Haemocomplettan® P/RiaSTAP(TM)
Number analyzed (Participants) | 21 | 21
h | 75.940 (23.831) | 69.378 (16.006)

12. Secondary Outcome: Mean Residence Time (MRT)
Description: as for outcome 3
Time Frame: Baseline to 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216, and 312 hours post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Octafibrin/FIBRYGA® | Haemocomplettan® P/RiaSTAP(TM)
Number analyzed (Participants) | 21 | 21
h | 106.272 (30.927) | 98.977 (20.812)

13. Secondary Outcome: Clearance
Description: as for outcome 3
Time Frame: Baseline to 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216, and 312 hours post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | Octafibrin/FIBRYGA® | Haemocomplettan® P/RiaSTAP(TM)
Number analyzed (Participants) | 21 | 21
mL/h/kg | 0.665 (0.197) | 0.804 (0.255)

14. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Description: as for outcome 3
Time Frame: Baseline to 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 216, and 312 hours post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Octafibrin/FIBRYGA® | Haemocomplettan® P/RiaSTAP(TM)
Number analyzed (Participants) | 21 | 21
mL/kg | 70.158 (29.860) | 76.631 (19.579)

ADVERSE EVENTS:
Description: Safety analysis dataset: All randomised participants who received at least 1 infusion of study medication (any part of an infusion of Octafibrin/FIBRYGA® and/or any part of an infusion of Haemocomplettan® P/RiaSTAP(TM)).
Arm/Group | Octafibrin/FIBRYGA® | Haemocomplettan® P/RiaSTAP(TM)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/22
Other Adverse Events (participants affected / at risk) | 11/22 | 11/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Octafibrin/FIBRYGA® (N=22) | Haemocomplettan® P/RiaSTAP(TM) (N=22)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Octafibrin/FIBRYGA® (N=22) | Haemocomplettan® P/RiaSTAP(TM) (N=22)
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 3
Mild allergic skin reaction (Immune system disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Octapharma agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Octapharma supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial. Octapharma also reserves the right to review data prior to publishing and provide comments/changes within a certain time period.